CLINICAL TRIAL: NCT04944407
Title: Minimal Invasive Laser Hemorrhoidoplasty vs Conventional Excisional Hemorrhoidectomy in II-III Grade Hemorrhoidal Disease: a Randomized Controlled Trial
Brief Title: Minimal Invasive Laser Hemorrhoidoplasty vs Conventional Excisional Hemorrhoidectomy in II-III Grade Hemorrhoidal Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Claudio Gambardella, Principal Investigator, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: laser hemorroid
Record Dates: First submitted 2021-06-15; First posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Hemorrhoids
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LHP GROUP (Experimental): patients recieved minimal invasive LHP procedure with diode laser
  Interventions: Procedure: LHP
- MM GROUP (Active Comparator): patients received conventional MM hemorroidectomy
  Interventions: Procedure: MM

INTERVENTIONS:
Procedure: LHP — A skin microincision of 3 mm was made about 1 to 1.5 cm of distance from the anal verge at the base of each hemorrhoidal node. The probe (1.85 mm of diameter) was driven through the incision in the submucosal tissue until reaching the area underneath the distal rectal mucosa. Then, ten to twelve effective pulses (adjusted to respective node dimensions), 8 watt per 3 seconds each, of approximately 24 Joule using a 1470-nm diode laser generator (LEONARDO® DUAL 45 Biolitec® Jena, Germany) were fired. Half of them were fired in the submucosal tissue, the others in the intra-nodal compartment determining the shrinkage of the hemorrhoidal piles. The anal wounds were left open. At the end of the procedure an anal tampon was positioned.
  Arms: LHP GROUP
Procedure: MM — The hemorrhoidectomy was performed by radiofrequency (LigaSure TM Small Jaw® Covidien®, Colorado, USA) or ultrasound (Focus® Ultracision® harmonic scalpel; Ethicon Endo-Surgery®, Inc., Cincinnati, Ohio). The anodermal wedge was incised, eventually removing external fibrosis and/or skin tags when present. Upward dissection started at this level with en-bloc excision of mucosal and submucosal layers from the underlying internal anal sphincter up to the anorectal ring. A compressive haemostatic sponge was left in place for 12-24 hours.
  Arms: MM GROUP

SUMMARY:
the study aims to evaluate the effectiveness and long term outcomes of laser hemorroidoplasty versus conventional milligan morgan hemorrhoidectomy in II-III degree hemorroidal disease.

DETAILED DESCRIPTION:
Background Hemorrhoidal disease (HD) is a widespread condition and several surgical techniques have been proposed to date without achieving a definitive consensus. Laser Hemorrhoidoplasty (LHP) is a minimal invasive procedure for HD treatment determining the shrinkage of the hemorrhoidal piles by diode laser limiting the postoperative discomfort and pain. The aim of the current prospective randomized trial is to evaluate the postoperative outcomes of HD patients undergoing LHP vs conventional Milligan-Morgan hemorrhoidectomy (MM).

Methods. Operative time, postoperative pain and complications, resolution of symptoms, patients 'quality of life, patients' evaluation of treatment and length of return to daily activity of II-III grade symptomatic HD patients undergoing LHP vs MM were prospectively evaluated. The patients were followed-up for 24 months looking for recurrence of prolapsed hemorrhoid or symptoms.

ELIGIBILITY:
Inclusion Criteria:

* II-III hemorrhoidal disease
* failure of conservative treatment
* ASA I-II

Exclusion Criteria:

* acutely thrombosed hemorrhoids
* patients affected by IBD involving rectum or anus
* patients previously surgically treated for hemorrhoidal disease and the inability to complete study protocol

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Pain evaluation | 30 postoperative days.
  postoperative pain assessment with Visual Analogue Scale Score
Analgesic use | 30 postoperative days.
  use of analgesic drugs in the postopertive days

SECONDARY OUTCOMES:
Presence of recurrence | 24 months
  Patients were considered to have recurrent hemorrhoidal symptoms when any of the following were recorded: bleeding, itching, pain or discomfort affecting patient's perception of quality of life, which could either be associated or not to prolapse recurrence. The Rovrik' score was adopted to assess this issue.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Campania Luigi Vanvitelli, Napoli, Italy

IPD SHARING:
Plan to Share IPD: Undecided
I am not sure in the current study phase